CLINICAL TRIAL: NCT05224115
Title: Biodistribution and Dosimetry in Human Healthy Volunteers of the Novel PET Radioligands [11C]CHDI-00485180-R and [11C]CHDI-00485626, Designed for Quantification of Cerebral Aggregated Mutant Huntingtin in Huntington's Disease.
Brief Title: Dosimetry of [11C]CHDI-180R and [11C]CHDI-626.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: s64086
Record Dates: First submitted 2022-01-13; First posted 2022-02-04 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Huntington Disease
Keywords: Positron Emission Tomography
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 2 urine samples for radio-activity assessments (3th sample prior to scanning for female participants for pregnancy test)
  * 6 venous blood samples for metabolite analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- [11C]CHDI-180R: Biodistribution and whole-body dosimetry for [11C]CHDI-00485180-R in 3 healthy volunteers.
  Interventions: Other: [11C]CHDI-00485180-R
- [11C]CHDI-626: Biodistribution and whole-body dosimetry for [11C]CHDI-00485626 in 3 healthy volunteers.
  Interventions: Other: [11C]CHDI-00485626

INTERVENTIONS:
Other: [11C]CHDI-00485180-R — Mutant huntingtin aggregate binding PET radioligand.
  Groups: [11C]CHDI-180R
Other: [11C]CHDI-00485626 — Mutant huntingtin aggregate binding PET radioligand.
  Groups: [11C]CHDI-626

SUMMARY:
A better understanding of the HD pathogenesis mechanisms may lead to a better understanding of disease pathology, progression and development of targeted therapies.

[11C]CHDI-00485180-R and [11C]CHDI-00485626 are two novel mutant huntingtin aggregate binding PET radioligands which have already demonstrated sensitivity to mutant huntingtin load in animal models. In the current study, the biodistribution and dosimetry of both these ligands will be investigated in young healthy volunteers according to a standard approach, in 3 subjects (including both genders) per tracer.

DETAILED DESCRIPTION:
For both groups, the dynamic whole-body distribution of the respective tracer labelled with [11C] will be measured after IV administration of 370 MBq. Two venous catheters, one on each arm, will be used for : 1/ the injection of [11C]CHDI-00485180-R or [11C]CHDI-00485626 tracer solution and 2/ for venous blood sampling (blood biochemistry and metabolites).

All images will be acquired using the SIEMENS Truepoint Biograph 40 PET-CT scanner. First, a CT scout will be acquired to set the axial field of view (FOV). The axial FOV should extend from the top of the head to the middle of the thighs (approximately 6-7 bed positions). Then, a low dose CT will be acquired for enabling PET attenuation correction and anatomical information (organ delineation). Following the CT, 10 sets of WB 3D PET images in total will be acquired sequentially. The first set of 9 whole body PET scans (scan segment 1) will be acquired, starting at the time of injecting [11C]CHDI-00485180-R solution or [11C]CHDI-00485626 solution. After this sequence of PET acquisitions, which will take up to 100 min, the subject will be moved out of the scanner and will be encouraged to void the bladder. After a 30 minute break, the subject will be repositioned in the PET/CT scanner and a second low dose CT will be acquired. WB scan 10 (scan segment 2) will be started at 2 hours after [11C]CHDI-00485180-R or [11C]CHDI-00485626 injection, scanning for a total scan duration of about 28 minutes.

During the first WB PET/CT scan segment, 6 venous blood samples (4 mL each) per subject will be taken at 5, 10, 20, 40, 60 and 100 min after [11C]CHDI-00485180-R or [11C]CHDI-00485626 injection. This will allow testing and further optimization of the HPLC metabolite analysis for future brain imaging studies with full kinetic modelling and quantification.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age between 18 and 55 years old
* Subject is judged to be in good health by the investigator on the basis of medical history. When still in doubt, a full physical and neurological examination can be conducted

Exclusion Criteria:

* Subject has a history of major internal disease that may interfere with the investigations (especially liver and kidney disease, cancer or uncontrolled diabetes).
* Subject has any history of a major neurological or psychiatric disorder
* Subject is currently smoker (> 20 cigarettes or equivalent/day) a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse.
* Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months.
* Subject suffers from claustrophobia or cannot tolerate confinement during PET-CT scanning procedures; subject cannot lie still for 90 minutes inside the scanner.
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e. weight lifting, running, bicycling) 3 days before and during the day of scanning.
* Subject does not understand the study procedure
* Subject is unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator.
* Subject is potentially pregnant (hCG will be performed in women with childbearing potential).
* Allergy for local anesthesia (lidocaine)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 6 young (18-55 years), healthy subjects, 3 for panel A ([11C]CHDI-00485180-R) and 3 for panel B [(11C]CHDI-00485626). Each panel should include both genders (i.e., 2M/1F or 2F/1M).
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Normalized cumulated activity coefficients (NCA) | Single point measure - during the acquisition of the PET scan (+- 2 hours 30minutes)
  Normalized cumulated activity coefficients (MBq-hr/hr) for indicated source organs determined from whole-body imaging.
Total organ doses | Single point measure - during the acquisition of the PET scan (+- 2 hours 30minutes)
  Total organ doses (µGy/MBq) for indicated target organs.
Effective doses (ED) | Single point measure - during the acquisition of the PET scan (+- 2 hours 30minutes)
  Effective doses (µSv/MBq) for indicated target organs.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Laere, MD, PhD, DSc, Principal Investigator — UZ/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delva A, Koole M, Serdons K, Bormans G, Liu L, Bard J, Khetarpal V, Dominguez C, Munoz-Sanjuan I, Wood A, Skinbjerg M, Wang Y, Vandenberghe W, Van Laere K. Biodistribution and dosimetry in human healthy volunteers of the PET radioligands [11C]CHDI-00485180-R and [11C]CHDI-00485626, designed for quantification of cerebral aggregated mutant huntingtin. Eur J Nucl Med Mol Imaging. 2022 Dec;50(1):48-60. doi: 10.1007/s00259-022-05945-z. Epub 2022 Aug 24. PMID 36001116
- See also: CHDI foundation — https://chdifoundation.org/